CLINICAL TRIAL: NCT07114666
Title: Efficacy and Safety of XH001 (New Antigen Tumor Vaccine) Combined With Chemotherapy as Adjuvant Therapy in Pancreatic Cancer Patients
Brief Title: XH001 (New Antigen Tumor Vaccine) Combined With Chemotherapy as Adjuvant Therapy in Pancreatic Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-25PJ0773
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XH001 (dose 1) (Experimental): Biological: XH001
  * mRNA neoantigen cancer vaccine（Dose 1） Drug: Chemotherapy
  * gemcitabine+capecitabine
  * oxaliplatin+lrinotecan+calcium folinate+5-FU
  Interventions: Biological: XH001; Drug: Chemotherapy
- XH001 (dose 2) (Experimental): Biological: XH001
  * mRNA neoantigen cancer vaccine(Dose 2) Drug: Chemotherapy
  * gemcitabine+capecitabine
  * oxaliplatin+lrinotecan+calcium folinate+5-FU
  Interventions: Biological: XH001; Drug: Chemotherapy

INTERVENTIONS:
Biological: XH001 — mRNA neoantigen cancer vaccine
Drug: Chemotherapy — Gemcitabine+Capecitabine or Oxaliplatin+lrinotecan+Calcium folinate+5-FU

SUMMARY:
This is a single-center, open label, single-arm, investigator-initiated study to evaluate the efficacy and safety of XH001 (neoantigen cancer vaccine) in combination with chemotherapy as Adjuvant Therapy in pancreatic cancer patients following surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form;
* Aged 18 to 75 years old;
* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma;
* R0 or R1 surgical resection as determined by pathology；
* Have not received any prior neoadjuvant therapy;
* ECOG score is 0 or 1;
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.

Exclusion Criteria:

* Borderline resectable pancreatic cancer;
* Evidence of metastasis or disease recurrence following surgical resection at any time;
* Evidence of malignant ascites;
* Pre-existing inflammatory bowel disease or the presence of complete or partial bowel obstruction, or persistent severe diarrhea after surgery;
* Needs to receive long-term systemic anti-allergic drug or known hypersensitivity to any component of the study treatment;
* History of autoimmune disease;
* Cerebrovascular accident (including ischemic stroke, hemorrhagic stroke, and transient ischemic attack) within 6 months before screening;
* Acute myocardial infarction within 6 months before screening, or uncontrolled angina, uncontrolled arrhythmia, severe heart failure (see Appendix 3, New York Heart Association Heart Failure Classification Criteria NYHA Class ≥ III) and other cardiovascular diseases;
* Received immunomodulatory medications within 4 weeks prior to the date of the first dose (D1) of XH001, including but not limited to: IL-2, CTLA-4 inhibitors, CD40 agonists, CD137 agonists, IFN-α;
* Received blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 7 days prior to the first dose of XH001;
* Received therapeutic tumor vaccines;
* With congenital or acquired immunodeficiency;
* Participating in other clinical trials and not enrolled at the screening period;
* Unable or unwilling to comply with the study protocol due to potential health, mental or social conditions in the opinion of the investigator;
* Other conditions that, in the opinion of the investigator, would make participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
DFS | From operation up to 36 months
  Disease Free Survival
DFS Rate | 12,24 and 36 months
  Disease-free survival rate
MFS | up to 36 months
  metastasis-free survival
OS | up to 48 months
  Overall survival

SECONDARY OUTCOMES:
Specific immune response | up to 36 months
  Antigen-specific T-cell responses
Adverse Event | up to 36 months
  Incidence and severity of adverse events (AEs), clinically significant abnormal changes in laboratory tests and other examinations (based on the Criteria for the Evaluation of Adverse Events [CTCAE] v5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rojas LA, Sethna Z, Soares KC, Olcese C, Pang N, Patterson E, Lihm J, Ceglia N, Guasp P, Chu A, Yu R, Chandra AK, Waters T, Ruan J, Amisaki M, Zebboudj A, Odgerel Z, Payne G, Derhovanessian E, Muller F, Rhee I, Yadav M, Dobrin A, Sadelain M, Luksza M, Cohen N, Tang L, Basturk O, Gonen M, Katz S, Do RK, Epstein AS, Momtaz P, Park W, Sugarman R, Varghese AM, Won E, Desai A, Wei AC, D'Angelica MI, Kingham TP, Mellman I, Merghoub T, Wolchok JD, Sahin U, Tureci O, Greenbaum BD, Jarnagin WR, Drebin J, O'Reilly EM, Balachandran VP. Personalized RNA neoantigen vaccines stimulate T cells in pancreatic cancer. Nature. 2023 Jun;618(7963):144-150. doi: 10.1038/s41586-023-06063-y. Epub 2023 May 10. PMID 37165196